CLINICAL TRIAL: NCT05586035
Title: Analysis of Factors and Treatment Related to Chronic Cough After Pulmonary Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: The People's Hospital of Gaozhou (Other); Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-Q-2022-007
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Persistent Cough; Pneumonectomy; Lung Neoplasms
MeSH Terms: conditions — Chronic Cough; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical resection is the primary treatment for pulmonary tumors. Surgeons has been frequently concerned about effectiveness, safety, and minimal invasive techniques. However, persistent cough, one of the most common complications of lung surgery, has received insufficient attention. This study set out to investigate the risk factors and treatment related to persistent cough after pulmonary resection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received pulmonary resection;
2. 18-to 85-year-old;
3. Pathologically diagnosed as NSCLC or benign tumor.

Exclusion Criteria:

1. Multiple malignancy in other parts of body;
2. Refuse to participate in this study;
3. Other situations evaluated by investigators not meet the enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients underwent pulmonary resection in Guangdong Provincial People's Hospital and Shenzhen People's Hospital were eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Occurence rate of persistent cough after pulmonary resection | Persistent cough after pulmonary resection is monitored from the time of surgery, up to 12 months.
  Occurence rate of persistent cough after pulmonary resection

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China